CLINICAL TRIAL: NCT01266616
Title: A Phase I Randomized, Partially Double-Blind, Placebo-Controlled, Dose-Escalation Study to Evaluate the Safety and Immunogenicity of a Cytokine Enhanced HIV-1 Multi-Antigen (HIV MAG) pDNA Vaccine Delivered Intramuscularly Followed by in Vivo Electroporation (IM/EP) or Intramuscularly in HIV-1 Infected Adults Receiving ART
Brief Title: Safety of and Immune Response to an Investigational HIV-1 Vaccine With or Without Interleukin-12 (IL-12) in HIV-1 Infected Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A5281; 10846 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 2010-12-23; First posted 2010-12-24 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Interleukin-12; Electroporation; HIV Therapeutic Vaccine
MeSH Terms: conditions — HIV Infections | interventions — Interleukin-12

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (10):
- Cohort 1: Vaccine alone IM/EP (Experimental): HIV MAG pDNA alone IM/EP
  Interventions: Biological: Profectus HIV MAG pDNA vaccine
- Cohort 1: Placebo (Placebo Comparator): Placebo given as an injection in each upper arm
  Interventions: Other: Placebo
- Cohort 2: Vaccine plus IL-12 IM/EP (Experimental): HIV MAG pDNA plus 50 mcg of IL-12 pDNA IM/EP
  Interventions: Biological: Profectus HIV MAG pDNA vaccine; Biological: IL-12
- Cohort 2: Placebo (Placebo Comparator): Placebo given as an injection in each upper arm
  Interventions: Other: Placebo
- Cohort 3: Vaccine plus IL-12 IM/EP (Experimental): HIV MAG pDNA plus 250 mcg of IL-12 pDNA IM/EP
  Interventions: Biological: Profectus HIV MAG pDNA vaccine; Biological: IL-12
- Cohort 3: Placebo (Placebo Comparator): Placebo given as an injection in each upper arm
  Interventions: Other: Placebo
- Cohort 4: Vaccine plus IL-12 IM/EP (Experimental): HIV MAG pDNA plus 1,000 mcg of IL-12 pDNA IM/EP
  Interventions: Biological: Profectus HIV MAG pDNA vaccine; Biological: IL-12
- Cohort 4: Placebo (Placebo Comparator): Placebo given as an injection in each upper arm
  Interventions: Other: Placebo
- Cohort 5: Vaccine plus IL-12 IM (Experimental): HIV MAG pDNA plus 1,000 mcg (or highest dose reached) IL-12 pDNA IM
  Interventions: Biological: Profectus HIV MAG pDNA vaccine; Biological: IL-12
- Cohort 5: Placebo (Placebo Comparator): Placebo given as an injection in each upper arm
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Profectus HIV MAG pDNA vaccine — 3,000 mcg admixture of two vaccine plasmids: ProfectusVax DNA Plasmid (HIV-1 gag/pol) and ProfectusVax DNA Plasmid (HIV-1 nef/tat/vif, env) at Weeks 0, 4, and 12
  Arms: Cohort 1: Vaccine alone IM/EP; Cohort 2: Vaccine plus IL-12 IM/EP; Cohort 3: Vaccine plus IL-12 IM/EP; Cohort 4: Vaccine plus IL-12 IM/EP; Cohort 5: Vaccine plus IL-12 IM
Biological: IL-12 — Administered at Weeks 0, 4, and 12
  Arms: Cohort 2: Vaccine plus IL-12 IM/EP; Cohort 3: Vaccine plus IL-12 IM/EP; Cohort 4: Vaccine plus IL-12 IM/EP; Cohort 5: Vaccine plus IL-12 IM
Other: Placebo — Saline injections at Weeks 0, 4, and 12
  Arms: Cohort 1: Placebo; Cohort 2: Placebo; Cohort 3: Placebo; Cohort 4: Placebo; Cohort 5: Placebo

SUMMARY:
Therapeutic HIV vaccines are designed to control HIV infection by boosting the body's natural immune response. There are currently no FDA-approved therapeutic HIV vaccines. This study will test whether giving an HIV-1 vaccine together with or without interleukin 12 (IL-12) is safe and effective. This study will also test a new way of giving the vaccine called electroporation (EP).

DETAILED DESCRIPTION:
Although highly active antiretroviral therapy (HAART) has greatly reduced HIV infection-related morbidity and mortality, individual response to therapy can be variable. Therapeutic vaccination works by augmenting virus-specific immunity and can be given with or without immunomodulatory agents or adjuvants. In conjunction with HAART, therapeutic vaccination may be a more effective treatment for the suppression of HIV-1 replication. This study will examine the safety and efficacy of giving an investigational vaccine with or without IL-12 in HIV-1 infected adults receiving HAART. This study will also test whether delivering the vaccine using EP is safe and increases the efficacy of the vaccine.

Participation in this study will last approximately 36 weeks. Participants will be randomly assigned to one of five cohorts. Cohort 1 will receive the HIV multi-antigen plasmid DNA (HIV MAG pDNA) vaccine or placebo intramuscularly (IM) in the upper arm followed by EP. Cohorts 2 through 4 will receive the HIV MAG pDNA vaccine and sequentially increasing doses of GENEVAX IL-12 pDNA or placebo by IM/EP. Cohort 5 will receive the HIV MAG pDNA vaccine with the highest dose of IL-12 pDNA or placebo by needle and syringe in the upper arm.

Participants receive two injections at Weeks 0, 4, and 12. Participants will complete a questionnaire that assesses the acceptability of the vaccine and remain at the clinic 30 minutes for observation after each vaccination. Participants will be contacted by telephone 2 to 3 days post-vaccination to assess vaccination-related signs and/or symptoms. All participants will be asked to record their temperatures and any symptoms they experience daily for 4 days following each vaccination on a Vaccination Report Card (VRC). All nonstudy vaccines or medications should also be recorded on the VRC. Study visits will occur at Weeks 0, 1, 2, 4, 5, 6, 8, 12, 13, 14, 16, 24, and 36. At most visits, participants will undergo a physical examination. Women of reproductive potential will also undergo pregnancy testing before receiving injections on Weeks 0, 4, and 12. Blood will be drawn at various time points to evaluate participants' health and measure immunologic markers, CD4 and CD8 T-cell counts, and cytokine levels. Blood and plasma will also be stored for future exploratory studies.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infected
* Stable antiretroviral therapy (ART) for a minimum of 6 consecutive months prior to study entry and intention to remain on stable ART until study completion
* CD4 T-cell count greater than or equal to 500 cells/mm3 (within 30 days prior to study entry)
* At least two measurements of HIV-1 RNA levels less than or equal to 200 copies/mL (first measurement must be performed at least 6 months prior to study entry and second measurement must be performed between 6 months prior to study entry and at least 30 days prior to study entry)
* Screening HIV-1 RNA less than 50 copies/mL (within 30 days prior to study entry)
* Hepatitis B surface antigen negative (within 30 days prior to study entry)
* Hepatitis C antibody negative or, if hepatitis C antibody positive, hepatitis C virus RNA negative (within 30 days prior to study entry)
* Certain laboratory values obtained within 30 days prior to study entry; more information can be found in the protocol
* Females of reproductive potential must have a negative urine pregnancy test within 3 days prior to study entry
* All study participants participating in sexual activity that could lead to pregnancy must agree to use at least one of the following forms of birth control for at least 21 days prior to study entry until the final study visit:

  * Condoms (male or female) with or without a spermicidal agent
  * Diaphragm or cervical cap with spermicide
  * Intrauterine device (IUD)
  * Hormone-based contraceptive
* Females who are not of reproductive potential are eligible without requiring the use of a contraceptive
* Ability and willingness of subject to provide written informed consent
* Collection of a pre-entry PBMC specimen for immunologic assays and entered into the Laboratory Data Management System (LDMS)

Exclusion Criteria:

* Confirmed (defined as two consecutive values) CD4 T-cell count less than 200 cells/mm3 at any time or any history or subject recollection of CD4 T-cell count less than 200 cells/mm3 prior to screening
* Any active malignancy that may require chemotherapy or radiation therapy
* Bleeding diathesis or condition associated with prolonged bleeding time that would contraindicate IM injection
* A skin-fold measurement of the cutaneous and subcutaneous tissue for eligible injection sites (on the medial deltoid muscles) that exceeds 40 mm
* Use of immunomodulatory, cytokine, or growth stimulating factors such as systemic corticosteroids, cyclosporine, methotrexate, azathioprine, anti-CD25 antibody, granulocyte macrophage colony-stimulating factor (GM-CSF), chondrocyte colony-stimulating factor (C-CSF), IFN, or interleukin-2 (IL-2) (within 30 days prior to study entry)
* Pregnancy or breastfeeding
* Use of any prior HIV vaccine (prophylactic and/or therapeutic) within 1 year before study entry
* Use of any investigational treatment within 6 months before study entry
* Use of any licensed or experimental non-HIV vaccination (e.g., hepatitis B, influenza, pneumococcal polysaccharide) within 4 weeks prior to study entry
* Use of any infusion blood product or immune globulin within 3 months prior to study entry
* Known or suspected hypersensitivity to any vaccine component, including hypersensitivity to amide-type local anesthetics, such as lidocaine (Xylocaine), mepivacaine (Polocaine/Carbocaine), etidocaine (Duranest), bupivacaine (Marcaine), or prilocaine
* Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements
* Serious illness requiring systemic treatment and/or hospitalization within 7 days prior to study entry
* Current use of any electronic stimulation device, such as cardiac demand pacemakers, automatic implantable cardiac defibrillators, nerve stimulators, or deep brain stimulators
* History of cardiac arrhythmia or palpitations (e.g., supraventricular tachycardia, atrial fibrillation, frequent ectopy, or sinus bradycardia [i.e., <50 beats per minute on exam]) prior to study entry (NOTE: Sinus arrhythmia is not excluded)
* History of syncope or fainting episode within 1 year of study entry
* Seizure disorder or any history of prior seizure
* Extensive tattoos covering the site of administration (upper left and right medial deltoid muscles)
* Presence of any surgical or traumatic metal implants at the site of administration (medial deltoid muscles)
* Any chronic inflammatory disease (e.g., ankylosing spondylitis, psoriasis, inflammatory bowel disease)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2011-03; Primary Completion 2012-10 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Occurrence of at least one greater than Grade 3 adverse event (AE) including signs/symptoms, lab toxicities, and/or clinical events that is possibly, probably, or definitely related to study treatment, as judged by the core team | From the first day of study treatment until 28 days after the last study vaccine administration
Change in the number of interferon (IFN)-gamma generating (in response to gag) CD4 T cells/million peripheral blood mononuclear cells (PBMCs) as measured by intracellular cytokine staining (ICS) | From Baseline to Week 14

SECONDARY OUTCOMES:
Answering "no" to the question, "In your opinion, would this study's vaccination procedure be acceptable as part of a treatment for HIV, if it proved to be effective?" | From Week 0 to Week 36
Answering "no" to the question, "In your opinion, would this study's vaccination procedure be acceptable if it could contribute to increased scientific knowledge about how best to administer vaccines to prevent or treat infections?" | From Week 0 to Week 36
Premature treatment discontinuation for reasons related to study treatment or related to any real or perceived effect of study vaccination or its administration | From Week 0 to Week 36
Rated pain (for participants administered vaccine/placebo by the EP device) | When the device was placed on the skin and the vaccine/placebo was injected; at the time of the electrical stimulation and muscle contraction; and at 10 and 30 minutes after the procedure was completed at Weeks 0, 4, and 12
Changes from baseline and absolute values of multiple functions of CD4 and CD8 T cells in response to gag and other vaccine-coded antigens individually and in sum | At Week 8, Week 14, and possibly other time points depending on the first set of data in an ICS assay

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Jacobson, MD, Study Chair — Division of Infectious Diseases and HIV Medicine, Drexel University College of Medicine
Locations (13):
- United States (13):
  - UCLA CARE Center CRS, Los Angeles, California
  - Stanford AIDS Clinical Trials Unit CRS, Palo Alto, California
  - Ucsf Hiv/Aids Crs, San Francisco, California
  - University of Colorado Hospital CRS, Aurora, Colorado
  - Massachusetts General Hospital Clinical Research Site (MGH CRS) CRS, Boston, Massachusetts
  - Brigham and Women's Hospital Therapeutics Clinical Research Site (BWH TCRS) CRS, Boston, Massachusetts
  - Washington University Therapeutics (WT) CRS, St Louis, Missouri
  - Trillium Health ACTG CRS, Rochester, New York
  - Univ. of Rochester ACTG CRS, Rochester, New York
  - Cincinnati CRS, Cincinnati, Ohio
  - Penn Therapeutics Crs, Philadelphia, Pennsylvania
  - University of Pittsburgh CRS, Pittsburgh, Pennsylvania
  - Houston AIDS Research Team CRS, Houston, Texas

REFERENCES:
- [Background] Finzi D, Blankson J, Siliciano JD, Margolick JB, Chadwick K, Pierson T, Smith K, Lisziewicz J, Lori F, Flexner C, Quinn TC, Chaisson RE, Rosenberg E, Walker B, Gange S, Gallant J, Siliciano RF. Latent infection of CD4+ T cells provides a mechanism for lifelong persistence of HIV-1, even in patients on effective combination therapy. Nat Med. 1999 May;5(5):512-7. doi: 10.1038/8394. PMID 10229227
- [Background] Koup RA, Safrit JT, Cao Y, Andrews CA, McLeod G, Borkowsky W, Farthing C, Ho DD. Temporal association of cellular immune responses with the initial control of viremia in primary human immunodeficiency virus type 1 syndrome. J Virol. 1994 Jul;68(7):4650-5. doi: 10.1128/JVI.68.7.4650-4655.1994. PMID 8207839
- [Background] Luxembourg A, Evans CF, Hannaman D. Electroporation-based DNA immunisation: translation to the clinic. Expert Opin Biol Ther. 2007 Nov;7(11):1647-64. doi: 10.1517/14712598.7.11.1647. PMID 17961089
- [Derived] Jacobson JM, Zheng L, Wilson CC, Tebas P, Matining RM, Egan MA, Eldridge J, Landay AL, Clifford DB, Luetkemeyer AF, Tiu J, Martinez AL, Janik J, Spitz TA, Hural J, McElrath J, Frahm N; ACTG A5281 Protocol Team. The Safety and Immunogenicity of an Interleukin-12-Enhanced Multiantigen DNA Vaccine Delivered by Electroporation for the Treatment of HIV-1 Infection. J Acquir Immune Defic Syndr. 2016 Feb 1;71(2):163-71. doi: 10.1097/QAI.0000000000000830. PMID 26761518